CLINICAL TRIAL: NCT06290063
Title: Rocky Mountain Cannabis Research Center - Cannabidiol and Older Adult Cannabis Users: A Randomized, Placebo-Controlled Study
Brief Title: Cannabidiol and Older Adult Cannabis Users
Acronym: QUARTz
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-08-0138
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sleep; Anxiety; Depression; Pain
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full-Spectrum Hemp-Derived CBD (fsCBD) (Experimental): 8 weeks of use of a daily dose of cannabis (200mg CBD/4mg THC)
  Interventions: Drug: fsCBD Cannabidiol
- Broad-Spectrum Hemp-Derived CBD (bsCBD) (Experimental): 8 weeks of use of a daily dose of cannabis (200mg CBD)
  Interventions: Drug: bsCBD Cannabidiol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fsCBD Cannabidiol — Full Spectrum hemp-derived CBD (fsCBD; 200mg CBD/4mg THC) capsules produced by Ecofibre/Ananda Hemp will be used
  Arms: Full-Spectrum Hemp-Derived CBD (fsCBD)
Drug: bsCBD Cannabidiol — Broad spectrum hemp-derived CBD (bsCBD; 200mg CBD) capsules produced by Ecofibre/Ananda Hemp will be used
  Arms: Broad-Spectrum Hemp-Derived CBD (bsCBD)
Drug: Placebo — Placebo arm; capsules produced by Ecofibre/Ananda Hemp will be used
  Arms: Placebo

SUMMARY:
Cannabis use increased 10 fold among adults over the age of 65 between 2014 and 2016 but very little data exists on the extent of their harmful effects on health and behavior. The overarching goal of this project is to test a novel harm reduction strategy in which older individuals who seek to use cannabis for pain, anxiety or mood problems (depression/anxiety) will be randomly assigned to one of three conditions in an 8 week randomized controlled trial: hemp-derived CBD+THC, hemp-derived CBD-THC, or placebo. This work has the ability to directly inform individual choices regarding the use of cannabis products among older adults, and direct policy decisions regulating cannabis formulations on the legal market.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years of age
* Able to provide informed consent
* Must have used a cannabis product at least once with no negative effects
* Must not have been regularly using any cannabis products (<3x/month) in the last 6 months
* Female participants must be postmenopausal
* Liver function tests (Alanine transaminase (ALT) and
* Aspartate transaminase (AST)) must show levels no greater than 2x the upper normal limits for age
* Must be currently taking medication/s for pain, sleep, and/or mood

Exclusion Criteria:

* Blood alcohol level > 0 at screening (to sign consent form)
* Report of other drug use (cocaine, opiates, methamphetamine) in the past 90 days or fail urine screen for any of these drugs
* Past or current diagnosis, or family history of diagnosis of psychosis
* Current use of anti-epileptic medications (e.g. clobazam, sodium valproate)
* Current use of medications known to have major interactions with Epidiolex (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, and/or teriflunomide).
* Current use of antipsychotic medications
* Currently undergoing chemotherapy (to prevent drug interactions)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Motor Function | Baseline, 4 weeks, 8 weeks
  Activities-specific Balance Confidence Scale. Participants asked about confidence in completion of 16 daily tasks without losing balance or becoming unsteady. Responses are on a scale from no confidence to completely confident, with higher aggregate scores meaning higher subjective motor function.
Balance | Baseline, 4 weeks, 8 weeks
  Dynamic sway (balance) measured via an app on a standard smartphone which will be attached to the participant's waist using a Velcro strap.
Anxiety | Baseline, 4 weeks, 8 weeks
  Beck Anxiety Inventory. 21 question survey. Each question is answered from 0 (not at all) to 3 (severely), where higher scores suggest higher anxiety. Total scores are between 0-63, where anything above 36 suggest potentially concerning levels of anxiety.
Depression | Baseline, 4 weeks, 8 weeks
  Beck Depression Inventory. 21 question survey. Each question is answered from 0 (not at all) to 3 (severely), where higher scores suggest higher depression. Total scores are between 0-63, where anything above 40 suggest potentially concerning levels of depression.
Blood Cytokine Levels | Baseline, 4 weeks, 8 weeks
  Blood cytokine levels will be measured from biological samples. Includes blood levels of cytokine inflammatory markers (IL6, TNF-α, IL-β, and CRP)
Depression/Anxiety | Baseline, 4 weeks, 8 weeks
  Depression Anxiety Stress Scale - 21 Item (DASS-21). Scores are between 0 and 63, with higher scores indicating more negative emotional states.
Drug Effects | 4 weeks, 8 weeks
  Drug Effects Questionnaire (DEQ). Six questions about drug effects with possible answers of "not at all", "somewhat", and "extremely", where higher scores indicate higher drug effects.
Inhibitory Control | Baseline, 4 weeks, 8 weeks
  Flanker Inhibitory Control and Attention Task
Cognitive Function | Baseline, 4 weeks, 8 weeks
  Functional Assessment of Cognitive Function - Cognitive (FACT-Cog). Scores are transformed such that scores range from 0-132 and higher scores indicate a better quality of life/cognitive function.
Pain Intensity and Interference | Baseline, 4 Weeks, 8 Weeks
  Brief Pain Inventory - Short Form (BPI - SF). Measures pain levels, pain interference, and relief from medication, and includes diagrams for labeling pain.
Cognitive Ability | Baseline, 4 weeks, 8 weeks
  Digital Symbol Substitution Test (DSST) assesses global cognitive ability
Pain Intensity | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Intensity (7-day). Scores are between 1-5, with 1 being no pain and 5 being very severe. Assessed with 2 items as well as current pain.
Change in Condition | 4 weeks, 8 weeks
  Patient Global Impression of Change (PGIC). 7 point scale assessing subjective changes in participant's condition.
Sleep Disturbance | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance 4a. Scores are separated between the first question (sleep quality) and the remaining 7 questions. For the first question, scores are between 1 and 5, with 1 being very poor sleep quality and 5 being very good sleep quality. The remaining 7 questions are scored individually on a scale of 1--5; for some questions, higher scores mean less disturbance, and for others, a higher score means more disturbance.
Sleep-Related Impairment | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep-Related Impairment 4a. Scores are between 4 and 20, with higher scores indicating more sleep-related impairment
Memory | Baseline, 4 weeks, 8 weeks
  Rey auditory verbal learning test assesses verbal memory.

SECONDARY OUTCOMES:
Polypharmacy-Pain Medications | Baseline, 4 weeks, 8 weeks
  Use of pain medications
Polypharmacy-Psychiatric Medications | Baseline, 4 weeks, 8 weeks
  Use of psychiatric medications
Polypharmacy-Sleep Medications | Baseline, 4 weeks, 8 weeks
  Use of sleep medications
Strength and Endurance | Baseline, 4 weeks, 8 weeks
  Leg strength and endurance measured with 30-second chair stand task. Participants are asked to stand up from a chair as many times as possible for 30 seconds.
Sleep Quality | Baseline, 4 weeks, 8 weeks
  PSQI (Pittsburgh Sleep Quality Index) measures quality and patterns of sleep. Global scores range from 0-21 with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado at Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No